CLINICAL TRIAL: NCT00764062
Title: Randomized Controlled Trial Short Antibiotic Therapy (3-Day) Versus Long Antibiotic Therapy (7-Day) in Odontology-Stomatology: Impact on the Resistance of Oral Streptococci
Brief Title: Amoxicillin Susceptibility of Oral Streptococci After a 3-Day or a 7-Day Amoxicillin Therapy
Acronym: ODAMOX
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was stopped earlier than planned because of the slow accrual rate.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Valérie MILLUL, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P040408
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2008-10-01 (Estimated); Status verified 2008-09

CONDITIONS: Odontogenic Infection
Keywords: Amoxicillin; Drug resistance, microbial; Streptococcus; Surgery, oral
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 7-day amoxicillin treatment (1g per os twice daily)
  Interventions: Drug: Amoxicillin
- 2 (Active Comparator): 3-day amoxicillin (1g per os twice daily) + 4-day placebo treatment (1g per os twice daily)
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — Amoxicillin :drug

SUMMARY:
Antibiotic resistance is a worldwide problem closely linked to antibiotic consumption. To limit the risk to select resistant bacteria, the rules of prescription are to use high doses and short durations of treatment. The purpose of this study was to evaluate the interest to reduce amoxicillin treatment from 7 days to 3 days, in cases of odontogenic infection requiring the extraction of the tooth associated with amoxicillin monotherapy. The 3-day treatment will be compared to the classical 7-day treatment for clinical efficacy (pain, wound healing) and impact on the susceptibility of oral streptococci to amoxicillin.

DETAILED DESCRIPTION:
Amoxicillin treatment starts the day of the inclusion in the study (day 0). Dentists and participants were blinded to treatment assignment for the duration of the study. The infected tooth was extracted 2 days after the beginning of the antibiotic treatment, and the post-operative follow-up was done 1 week after tooth extraction (day 9). An additional follow-up was done one month later (day 30).

Clinical parameters were collected one week after tooth extraction (day 9). Pain was evaluated by its intensity during the days following surgery (using an analog visual scale varying from 0 -no pain- to 10 -very intense pain-), and by the total amount (in mg) of paracetamol ingested. The infectious state was evaluated by local wound healing, regional adenopathy and fever. The wound healing score combined local inflammation and sensitivity, and the presence or absence of a blood clot.

The streptococci resistance was assessed at the patient-level by the proportion of patient with at least one resistant streptococcus, and at the streptococcus-level by the proportion of resistant streptococcus out of the total streptococci flora. Intermediate susceptibility to amoxicillin was defined as a minimum inhibitory concentration (MIC) of 0.5-16 mg/L; resistance was defined as an MIC greater than or equal to 16 mg/L.

ELIGIBILITY:
Inclusion Criteria:

* odontogenic infection requiring tooth extraction asociated with amoxicillin monotherapy
* good condition
* 18-60 years old
* written informed consent provided

Exclusion Criteria:

* antibiotic prophylactic treatment
* special infectious risk (immunodeficiency, diabetes..)
* pregnant or breastfeeding women
* amoxicillin contraindication
* antibiotic treatment during the lasts 45 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2005-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Susceptibility to amoxicillin of oral streptococci | at day 0, day 9 and day 30.

SECONDARY OUTCOMES:
Non-inferiority of clinical efficacy | at day 9

CONTACTS AND LOCATIONS:
Overall Officials: Hélène CHARDIN, DD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Paris, France